CLINICAL TRIAL: NCT04782167
Title: Comparison Of Brace (Balance, Resistance, Aerobic, Cognitive Exercise) And Proprioceptive Training On Balance And Mobility In Knee Osteoarthritis
Brief Title: Proprioception and BRACE Training in Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: khadija liaquat (Other)
Responsible Party: Sponsor-Investigator, khadija liaquat, Senior Lecturer, Riphah International University
Organization: Riphah International University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Riphah IU Ali
Record Dates: First submitted 2021-03-01; First posted 2021-03-04 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Osteoarthritis Knees Both
Keywords: proprioception training, balance, BBS,
MeSH Terms: interventions — Braces

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Proprioception training (Experimental): Researcher give proprioception protocol to one group
  Interventions: Behavioral: Propirioceptive training
- Brace (Experimental): Researcher give BRace training to one group
  Interventions: Behavioral: BRACE

INTERVENTIONS:
Behavioral: BRACE — Balance training,Static balance:
  1. Romberg with eye open & eye close [30 sec repeat 3 times]
  2. Tandem standing with eye open then with eye close. Right foot front first, then left foot front [10 Sec repeat 3 times]
  3. Single leg stance 5 repetition with sec.
  Static/Dynamic/Anti-cipatory Postural Control:
  1. Sit to stand: 5 repetition
  2. Functional reach test: forward, sideways & cross reach, practice 1 min for each
  3. TUG test: with distance of 10 feet & time 10 sec. practice 2 min Cognitive exercises
  1) Count reverse from 50 Repeat with eyes open and close Reps of 30s for each 2) Push wall and reverse count from 20 3) Remember 5 words, Name 5 animals, Repeat 5 words
  Arms: Brace
Behavioral: Propirioceptive training — 1st Phase - Steady phase (1st set: Eyes Open, 2nd set: Eyes Close) Preserve standup position Equally heels up and down Preserve standup on one leg by turns
  Arms: Proprioception training

SUMMARY:
Knee osteoarthritis is common joint disorder in older adults. The prevalence of osteoarthritis is increasing in the elderly population and due to obesity.The aim of this study to compare improvement in balance between BRACE and proprioceptive training in knee osteoarthritis and to compare mobility level between proprioceptive and BRACE in knee osteoarthritis

DETAILED DESCRIPTION:
Knee osteoarthritis is common joint disorder in older adults. The prevalence of osteoarthritis is increasing in the elderly population and due to obesity. Balance disorder generally disturbed equilibrium and increase risk of fall. There is lack of proprioceptive sensation in patients with knee osteoarthritis. The aim of this study to compare improvement in balance between BRACE and proprioceptive training in knee osteoarthritis and to compare mobility level between proprioceptive and BRACE in knee osteoarthritis. Randomized control trial study of 8 week follows up. Sample size will be 22. The patients will be divided into 2 groups BRACE and proprioceptive training. The patients will get training section for 3 days per week for 8 weeks. The measurement will be taken at base line, after 8 weeks. Study duration will be 6 months. Individuals of age 50-70 year, Mini-mental state examination (MMSE) 20 or higher, Berg Balance Scale (BBS) 30-45 points, Experience of at least one fall during the previous 12 months, both Males and Females will be include. Patients will be excluded if they exhibited history of cardiovascular or musculoskeletal diseases, previously used medication for the central nervous system, occurrence of lower limbs lesions or fractures in last six months. Assessment tools will be MMSE, Berg balance scale, TUG, CTSIB, 6 minute walk test. Data will be analyzed through SPSS 20. Data will be check for its normality, within groups comparison paired sample T-test, between groups independent sample T-test will be used

ELIGIBILITY:
Inclusion Criteria:

* Age 50-70 years.
* Both Males and Females
* Knee osteoarthritis unilateral and bilateral (12).
* American College of Rheumatology (ACR) criteria for diagnosing osteoarthritis of knee joint is presence of pain in knee joint plus any three of six factors listed below (13).
* Age more than 50 y
* Presence of crepitus on active motion
* Less than 30 min of morning stiffness
* Bony tenderness
* Bony overgrowth
* No palpable warmth of synovium
* Mini-mental state examination (MMSE) 23 or higher (14).
* Berg Balance Scale (BBS) 30-45 points (4)

Exclusion Criteria:

* History of stroke during the previous 12 months
* History of cardiovascular or musculoskeletal diseases,

  * Previously used medication for the central nervous system.
* Presence of lower limb lesions or fractures in the last six months

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
Berg balance scale | 20 minutes
  it is measure of dynamic and static balance
Time up and go test | less than 3 minutes
  it is also measure of static and dynamic balance
clinical test of sensory interaction on balance | 20 minutes
  test for balance

CONTACTS AND LOCATIONS:
Locations (1):
- Independent University Hospital, faisalabad, Faisalābad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No